CLINICAL TRIAL: NCT03617887
Title: Isometric Abdominal and Specific Gluteus Medius Work in Soccer Players. A Randomized Pilot Study
Brief Title: Isometric Abdominal and Specific Gluteus Medius Work in Soccer Players
Acronym: COREGLUTFEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Real Fundación Victoria Eugenia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COREGLUTFEM
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Young Soccer Players
Keywords: Core; Isometric abdominal; Gluteus medius; Adductor; Lumbo-pelvic stability
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: 25 subjects will be randomized into both groups: experimental and control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Plank exercise, Lateral plank exercise, Bird dog exercise, Pelvic drop exercise, and Stabilization of the middle gluteus in the knee valgus:
  Interventions: Other: Experimental group
- Control group (Experimental): Plank exercise, Lateral plank exercise and Bird dog exercise
  Interventions: Other: Control group

INTERVENTIONS:
Other: Experimental group — Plank exercise, Lateral plank exercise, Bird dog exercise, Pelvic drop exercise, and Stabilization of the middle gluteus in the knee valgus.
  The intervention consisted of sessions of approximately 20 minutes, taking place 2 days a week, for 8 weeks. The exercises were performed at the beginning of the training session, and consisted of a work of the abdominal region in the control group, and a specific work of gluteus medius, added to the previous one, in the experimental group.
  Arms: Experimental group
Other: Control group — Plank exercise, Lateral plank exercise and Bird dog exercise. The intervention consisted of sessions of approximately 20 minutes, taking place 2 days a week, for 8 weeks. The exercises were performed at the beginning of the training session, and consisted of a work of the abdominal region.
  Arms: Control group

SUMMARY:
The problems of lack of lumbo-pelvic stability, as well as weakness or mobile restriction of the adductor muscles, may be the origin of lower limb injuries. Both intrinsic and extrinsic factors are key in the probability of suffering an imbalance. A protocol of abdominal isometric strength, accompanied by specific exercises of the gluteus medius, can be useful in order to prevent such dysfunctions.

The objective is to compare the efficacy of abdominal isometric work against the specific work of gluteus medius in the improvement of lumbo-pelvic stability and strength and elasticity of the adductor muscles.

Study design. Randomized, longitudinal, experimental, prospective, multicentre and single-blind clinical trial. It will take place at the facilities of the Soccer Club Fuenlabrada S. A. D. and the European University of Madrid.

The subjects will be randomly divided into two groups: control group and experimental group. The intervention period will last eight weeks, performing 2 weekly sessions, of approximately 20 minutes (depending on the group to which each subject belongs). The variables to be evaluated before and after the intervention will be the lumbo-pelvic stability and the strength and elasticity of the adductor muscles. For the statistical analysis, the SPSS program version 19.0 will be used.

It is expected to find how gluteal work produces improvements in lumbo-pelvic stability, as well as an increase in strength and adduction elasticity.

DETAILED DESCRIPTION:
Each session will last 20 minutes, taking place during 2 days a week, in a period of 8 weeks. The intervention will be carried out at the beginning of the training session. This intervention consists of an abdominal work protocol, and a gluteal work protocol added to the previous protocol, performed by the control group and the experimental group, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years
* Federated in the Royal Football Federation of Madrid currently and with a minimum of 4 years
* Without any previous pathology or during the experimental period
* Signed the informed consent

Exclusion Criteria:

* Not have current or previous pathology in any region of the lower limb during the last 6 months
* Inability or inability to comply with the demands of the study in terms of follow-up or problems of involvement
* Players under pharmacological treatment or exercising a physiotherapy treatment parallel to the development of the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline lumbo-pelvic stability after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  With a universal goniometer, the subject slightly lowers the extended legs, and the moment the lumbar spine loses contact with the ground, the angle is measured whose legs form with the ground

SECONDARY OUTCOMES:
Change from baseline elasticity of the adductor muscles after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  With the subject sitting on the floor, and both legs extended and separated as much as possible, passively, place the goniometer with the axis parallel to the floor at the level of the pubic symphysis and both arms moving along the axis of the femur. The normative values: the normal range is from 0º to 180º
Change from baseline adductor muscle strength after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  With a manual dynamometer, hooked to a fixed point and perpendicular and lateral to the leg to be treated, at the height of the distal third of the tibia, and the subject standing, the subject had to perform a hip adduction, generating a Progressive maximum isometric contraction.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Royal Victoria Eugenia Foundation, Madrid, Madird, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guerrero-Tapia H, Martin-Baeza R, Cuesta-Barriuso R. Effectiveness of Abdominal and Gluteus Medius Training in Lumbo-Pelvic Stability and Adductor Strength in Female Soccer Players. A Randomized Controlled Study. Int J Environ Res Public Health. 2021 Feb 5;18(4):1528. doi: 10.3390/ijerph18041528. PMID 33562743